CLINICAL TRIAL: NCT01521234
Title: Using Wireless Technology in Clinical Practice: Does Feedback of Daily Walking Activity Improve Walking Outcomes of Individuals Receiving Rehabilitation Post-stroke?
Brief Title: Using Wireless-technology for Feedback of Daily Walking Activity Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Avril Mansfield, Post-doctoral fellow, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OSN-Mansfield-2011
Record Dates: First submitted 2012-01-23; First posted 2012-01-30 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback group (Experimental): For participants assigned to the feedback group, physiotherapists will receive a summary of patients' walking activity for the previous week as a tool to guide goal planning. Physiotherapists will use the information as a 'homework checker' to determine if patients are complying with an assigned walking program. In the case of non-compliance, the physiotherapist will discuss a coping strategy for better integrating walking activity into the patients' day. In the event that the patient is meeting their specific sub-goals for walking activity, the physiotherapist will re-evaluate these sub-goals and suggest more challenging goals.
  Interventions: Behavioral: Feedback of daily walking activity
- No-feedback group (No Intervention): For participants assigned to the control group, physiotherapists will not receive accelerometer-based feedback of daily walking activity. However, physiotherapists will still discuss the achievement of walking goals with their patients. This is usual care around goal planning.

INTERVENTIONS:
Behavioral: Feedback of daily walking activity — Participants will wear accelerometers every weekday during in-patient rehabilitation to monitor walking activity. Feedback of daily walking activity will be provided to the patients' treating physiotherapists to assist with goal-planning around walking.
  Arms: Feedback group

SUMMARY:
Regaining independent walking is the top priority for individuals recovering from stroke. Thus, physical rehabilitation post-stroke should focus on improving walking function and endurance. However, the amount of walking completed by individuals with stroke attending rehabilitation is far below that required for independent community ambulation. There has been increased interest in accelerometer-based monitoring of walking post-stroke. Walking monitoring could be integrated within the goal-setting process for those with ambulation goals in rehabilitation. The purpose of this study is to determine the effect of accelerometer-based feedback of daily walking activity during rehabilitation on the frequency and duration of walking post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* individuals with sub-acute stroke attending in-patient rehabilitation at Toronto Rehab
* patients who have identified improving walking function as a rehabilitation goal
* patients who can walk without supervision at the time of recruitment into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in walking activity from admission to discharge from rehabilitation | Admission and discharge from in-patient rehabilitation (approx. 4-6 weeks)
  Total daily walking acitivty, measured by number of steps per day, total duration of walking activity, total distance walked, and frequency of 'long' walking bouts (>5 minutes in duration).
Change in control of walking | Admission and discharge from in-patient rehabilitation (approx. 4-6 weeks)
  Self-selected walking speed and symmetry of spatio-temporal characteristics of walking

SECONDARY OUTCOMES:
Change in self-efficacy | Admission and discharge from in-patient rehabilitation (approx. 4-6 weeks)
  Stroke self-efficacy questionnaire
Goal attainment | Discharge from in-patient rehabilitation (4-6 weeks), discharge from out-patient rehabilitation (10-16 weeks)
  Rehabilitation goals are classified as 'achieved', 'partially achieved', 'not completed' or 'discontinued'.
Community integration | Discharge from out-patient rehabilitation (10-16 weeks) and 3-month follow-up
  Community integration questionnaire
Satisfaction with progress towards rehabilitation goals | Discharge from in-patient rehabilitation (4-6 weeks) and discharge from out-patient rehabilitation (10-16 weeks)
  Participants will be asked to rate satisfaction with progress towards goals on a 10-point scale
Barriers to walking | Monitored throughout participants' enrolment (0-28 weeks)
  Open-ended question regarding participants' perceived barriers to walking.
Falls | Monitored throughout participants' enrolment (0-28 weeks)
  Increased walking activity might increase the risk for falls. Falls experienced throughout the study will be recorded to determine if there are more falls in the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Avril Mansfield, PhD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- [Background] Prajapati SK, Gage WH, Brooks D, Black SE, McIlroy WE. A novel approach to ambulatory monitoring: investigation into the quantity and control of everyday walking in patients with subacute stroke. Neurorehabil Neural Repair. 2011 Jan;25(1):6-14. doi: 10.1177/1545968310374189. Epub 2010 Sep 9. PMID 20829413
- [Background] Mansfield A, Wong JS, Bayley M, Biasin L, Brooks D, Brunton K, Howe JA, Inness EL, Jones S, Lymburner J, Mileris R, McIlroy WE. Using wireless technology in clinical practice: does feedback of daily walking activity improve walking outcomes of individuals receiving rehabilitation post-stroke? Study protocol for a randomized controlled trial. BMC Neurol. 2013 Jul 18;13:93. doi: 10.1186/1471-2377-13-93. PMID 23865593
- [Result] Mansfield A, Wong JS, Bryce J, Brunton K, Inness EL, Knorr S, Jones S, Taati B, McIlroy WE. Use of Accelerometer-Based Feedback of Walking Activity for Appraising Progress With Walking-Related Goals in Inpatient Stroke Rehabilitation: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2015 Oct;29(9):847-57. doi: 10.1177/1545968314567968. Epub 2015 Jan 20. PMID 25605632